CLINICAL TRIAL: NCT01698554
Title: Bimatoprost in the Treatment of Eyelash Hypotrichosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-046; 2012-003007-35 (EudraCT Number)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Idiopathic Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- bimatoprost formulation A solution (Experimental): Bimatoprost formulation A solution single-dose vial applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Interventions: Drug: bimatoprost formulation A solution
- bimatoprost solution 0.03 % (Active Comparator): Bimatoprost solution 0.03 % (LATISSE®) multi-dose vial applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Interventions: Drug: bimatoprost solution 0.03 %
- vehicle of bimatoprost formulation A solution (Placebo Comparator): Vehicle of bimatoprost formulation A solution single-dose vial applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Interventions: Drug: vehicle of bimatoprost formulation A solution
- vehicle of bimatoprost solution 0.03 % (Placebo Comparator): Vehicle of bimatoprost solution 0.03 % multi-dose vial applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Interventions: Drug: vehicle of bimatoprost solution 0.03 %

INTERVENTIONS:
Drug: bimatoprost formulation A solution — Bimatoprost formulation A solution applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Arms: bimatoprost formulation A solution
Drug: bimatoprost solution 0.03 % — Bimatoprost solution 0.03 % (LATISSE®) applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Other Names: LATISSE®
  Arms: bimatoprost solution 0.03 %
Drug: vehicle of bimatoprost formulation A solution — Vehicle of bimatoprost formulation A solution applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Arms: vehicle of bimatoprost formulation A solution
Drug: vehicle of bimatoprost solution 0.03 % — Vehicle of bimatoprost solution 0.03 % applied to the upper eyelid of both eyes once daily for 4 months using the supplied applicator.
  Arms: vehicle of bimatoprost solution 0.03 %

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost solution formulation A compared with bimatoprost solution 0.03% (LATISSE®) and vehicle in the treatment of eyelash hypotrichosis (inadequate eyelashes).

ELIGIBILITY:
Inclusion Criteria:

-Male and female adult patients with eyelash hypotrichosis (inadequate eyelash growth).

Exclusion Criteria:

* Damage to eyelid area (scarring) that may prevent growth of eyelashes
* Active eye diseases (glaucoma, uveitis, eye infections, chronic blepharitis or severe dry eye)
* Eye or eyelid surgery (including laser, refractive, intraocular filtering surgery, blepharoplasty) during the 3 months prior to screening
* Current eyelash implants of any kind
* Eyelash tint or dye application within 2 months of baseline
* Eyelash extensions application within 3 months of baseline
* Use of eyelash growth products within 6 months of baseline
* Treatments that may affect hair growth (minoxidil, cancer chemotherapeutic agents, etc) within 6 months prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Newport Beach, California, United States
- Saint Petersburg, Russia
- Stockholm, Sweden
- Norfolk, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Started | 153 | 157 | 75 | 79
Completed | 147 | 147 | 73 | 77
Not Completed | 6 | 10 | 2 | 2
Not completed — Adverse Event | 2 | 5 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Personal Reasons | 0 | 5 | 1 | 1
Not completed — Protocol Violation | 2 | 0 | 1 | 0
Not completed — Other Miscellaneous Reasons | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 % | Total
Number analyzed (Participants) | 153 | 157 | 75 | 79 | 464
Age, Customized [Number; unit: Participants]
  <45 years | 27 | 34 | 16 | 15 | 92
  45 to 65 years | 104 | 106 | 47 | 55 | 312
  >65 years | 22 | 17 | 12 | 9 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 153 | 75 | 79 | 457
  Male | 3 | 4 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Grade Increase (Improvement) From Baseline in the Investigator's Assessment of Overall Eyelash Prominence (GEA)
Description: The investigator evaluated the overall eyelash prominence in both eyes using the GEA 4-point scale: 1= minimal, 2= moderate, 3= marked and 4= very marked. A 1-grade improvement in the GEA score from Baseline indicated improvement.
Time Frame: Baseline, Month 4
Population: Intent-to-treat (ITT) Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Number analyzed (Participants) | 153 | 157 | 75 | 79
percentage of participants | 82.4 | 83.4 | 24.0 | 20.3

2. Secondary Outcome: Change From Baseline in Upper Eyelash Length as Measured Using Digital Image Analysis (DIA)
Description: Photographs were taken of the eyelashes and assessed using DIA. Length was measured in millimeters (mm). Data from both eyes were averaged for each participant for analysis. A positive change from Baseline indicated longer length (improvement)
Time Frame: Baseline, Month 4
Population: Participants from the ITT Population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Number analyzed (Participants) | 152 | 157 | 75 | 79
mm
  Baseline | 6.09 (0.856) | 5.97 (0.789) | 5.90 (0.812) | 6.03 (0.852)
  Change from Baseline at Month 4 | 1.61 (0.888) | 1.62 (0.955) | 0.08 (0.442) | 0.05 (0.482)

3. Secondary Outcome: Change From Baseline in Upper Eyelash Thickness/Fullness as Measured Using DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash thickness (fullness) was measured in millimeters squared (mm^2). Data from both eyes were averaged for each participant for analysis. A positive change from Baseline indicated fuller eyelashes (improvement).
Time Frame: Baseline Month 4
Population: Participants from the ITT Population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Number analyzed (Participants) | 151 | 156 | 74 | 78
mm^2
  Baseline | 0.85 (0.400) | 0.82 (0.404) | 0.76 (0.333) | 0.81 (0.380)
  Change from Baseline At Month 4 | 0.58 (0.359) | 0.64 (0.392) | 0.02 (0.196) | 0.03 (0.237)

4. Secondary Outcome: Change From Baseline in Upper Eyelash Intensity (Darkness) as Measured Using DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash darkness (intensity) was measured in both eyes and averaged for analysis using a scale where 0=black and 255=white. A negative change from Baseline indicated darker eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the ITT Population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: intensity units
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Number analyzed (Participants) | 151 | 156 | 74 | 78
intensity units
  Baseline | 145.33 (24.024) | 147.39 (24.934) | 147.44 (22.323) | 145.79 (26.670)
  Change from Baseline at Month 4 | -23.98 (15.719) | -24.78 (16.417) | -2.78 (10.443) | 0.17 (10.065)

5. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied in the Patient's Assessment of Overall Eyelash Satisfaction as Measured by the Eyelash Satisfaction Questionnaire (ESQ-9)
Description: Participants rated their overall eyelash satisfaction by answering Eyelash Satisfaction Questionnaire (ESQ-9) question #3: "Overall, how satisfied are you with your eyelashes?" using a 5-point scale: 1= very unsatisfied (worst), 2= unsatisfied, 3= neutral, 4= satisfied or 5= very satisfied (best). The percentage of participants who rated their satisfaction as satisfied or very satisfied at Month 4 is reported.
Time Frame: Month 4
Population: ITT Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Number analyzed (Participants) | 153 | 157 | 75 | 79
percentage of participants | 71.2 | 65.0 | 28.0 | 20.3

ADVERSE EVENTS:
Arm/Group | Bimatoprost Formulation A Solution | Bimatoprost Solution 0.03 % | Vehicle of Bimatoprost Formulation A Solution | Vehicle of Bimatoprost Solution 0.03 %
Serious Adverse Events (participants affected / at risk) | 0/153 | 5/157 | 1/75 | 1/79
Other Adverse Events (participants affected / at risk) | 7/153 | 8/157 | 3/75 | 3/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bimatoprost Formulation A Solution (N=153) | Bimatoprost Solution 0.03 % (N=157) | Vehicle of Bimatoprost Formulation A Solution (N=75) | Vehicle of Bimatoprost Solution 0.03 % (N=79)
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0/150 | 0/153 | 0 | 1 — female population
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Formulation A Solution (N=153) | Bimatoprost Solution 0.03 % (N=157) | Vehicle of Bimatoprost Formulation A Solution (N=75) | Vehicle of Bimatoprost Solution 0.03 % (N=79)
Intraocular pressure decreased (Investigations) | 7 | 8 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.